CLINICAL TRIAL: NCT00285831
Title: Dysphoric-like Disorder of Epilepsy, Is it Unique?
Brief Title: Mild Depression 2 Week Observational Study
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: GlaxoSmithKline (Industry); Long Island Jewish Medical Center (Other); Rush University Medical Center (Other)
Other Study IDs: 95879
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to assess whether the dysphoric-like depressive characteristics observed in people with epilepsy are unique to this patient population in comparison to three control groups: Mild Depression (enrolled at Stanford University), Migraine Headaches (enrolled at Long Island Jewish Medical Center), and Multiple Sclerosis (enrolled at Rush University Medical Center).

DETAILED DESCRIPTION:
This is a multicenter study consisting of a Screen and Retest phase conducted in two separate days separated by a two-week period. After providing written informed consent and meeting protocol-defined inclusion criteria at Screen, patients will be administered the Wide Range Achievement Test 3 (WRAT3) to ensure adequate word reading ability with which to complete the self-report forms. Patients who achieve a satisfactory score will be interviewed using the Mini International Neuropsychiatric Interview (MINI). Afterwards, each patient will first complete the 46 item Mood and Anxiety Symptom List in Epilepsy (MAS-E) and then five additional questionnaires in random order. Patients will also be given the opportunity to be rated by a proxy (e.g., caregiver, family member, friend) who will also complete the MAS-E.

Patients will return the completed documents to the investigator and be given an additional MAS-E to take home. In the Retest phase, patients will be asked to complete the MAS-E again exactly 14 days from the date of the Screen visit. The proxy will also be given an additional MAS-E and be asked to complete the MAS-E exactly 14 days from completion of the first MAS-E. The documents shall be returned to the clinic via U.S. mail on the same day of completion. It is not necessary to have a proxy to participate in this study.

Total study participation takes 2 weeks and approximately one visit to the clinic for the screening visit.

ELIGIBILITY:
Inclusion Criteria::

" Male or female 18 years of age or older. " Presence of a Depressive disorder that presents as a dysthymic or minor depressive disorder and whose score on the Beck Depression Inventory (BDI) range between 11 and 20. Patients with major depression will be excluded.

" Is currently on stable doses of medications i.e., no change in treatment in the previous 30 days.

" Achieves a satisfactory score on the WRAT3 (standard score is > 69). " Is capable of completing the self-reporting questionnaires. " Is willing and able to provide written informed consent and comply with the study protocol
 Exclusion Criteria:" Presence of a clinically significant comorbidity of an unstable or progressive nature (e.g., psychosis, delirium) that could, in the opinion of the investigator, prevent completion of the questionnaires or warrant immediate medical intervention.

" Participation in an investigational trial within the past 30 days. " Inability to communicate well with site study personnel, e.g. inability to read or understand English, poor mental development or impaired brain function.

" Patients with a clinical picture that meets criterion of major depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-12 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J Barry, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States